CLINICAL TRIAL: NCT05457335
Title: Shanghai First Maternity and Infant Hospital,
Brief Title: 2.Comparison of the Live Birth Rate of PGT Versus Expectant Management in Patients With RPL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, chen zhi qin, clinical doctor in chief, Shanghai First Maternity and Infant Hospital
Other Study IDs: shanghai first maternity
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Outcome; Time-to-Pregnancy
Keywords: preimplantation genetic testing; expectant management; live birth rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PGT-A group: For patients undergoing PGT-A, trophectoderm biopsy was performed on good quality blastocysts and about five cells were aspirated gently and separated from the blastocyst by applying multiple pulses of a noncontact 1.48- μm diode laser (Saturn 5 ActiveTM, Cooper Surgical, Inc., CT, USA) through a zona pellucida opening created by the laser. The biopsied cells were washed three times in 1 × phosphate buffered saline (PBS) (Life Technologies, NY, USA), transferred to a PCR tube containing 2.5 μl 1× PBS and cryopreserved at -80◦C until analysis. Genetic laboratories analyzed and interpreted biopsies. The genetic screening was performed using the next-generation sequencing (NGS)-based assay VeriSeq PGS following standard protocols and manufacturer recommendations (Illumina Inc., San Diego, USA）. The PGT-A report can be euploid, aneuploidy, mosaic and non-conclusive. Euploid embryos were transferred while aneuploid and mosaic embryos were not replaced.
  Interventions: Procedure: undergoing PGT
- Expectant management group: In the this group, one attempt at conception was defined as one calendar months trying to conceive spontaneously. Either in natural cycles for ovulatory women and in clomiphene/letrozol induced cycles for anovulatory women with or without ultrasound monitoring.
  Interventions: Procedure: undergoing PGT

INTERVENTIONS:
Procedure: undergoing PGT — Preimplantation genetic testing for aneuploidy

SUMMARY:
Recurrent pregnancy loss (RPL) is a multifactorial disorder defined by the American Society for Reproductive Medicine (ASRM) as two or more clinical miscarriages (CMs). However, US guidelines differ with European guidelines which defined recurrent miscarriage as three consecutive prior pregnancy losses (The Royal College of Obstetricians and Gynaecologists Green-Top Guideline, 2011). Thus, there is currently no uniformly agreed upon definition of RPL, the ASRM recommends that a clinical evaluation for RPL commence following two early pregnancy losses, and that a threshold of three prior pregnancy losses be utilized for epidemiologic studies (The Practice Committee of the American Society for Reproductive Medicine, 2012).

Although the overall incidence of RPL is low and estimated at 5% of women (The Practice Committee of the American Society for Reproductive Medicine, 2012), it presents a significant diagnostic and treatment challenge for both patients and clinicians. Guidelines for the evaluation of patients with RPL include evaluation of the uterine cavity and blood work to determine parental karyotypes and the presence of anti-phospholipid antibodies (APLA). In at least 50% of patients, however, an etiology for RPL is not identified (Stirrat, 1990; Stephenson, 1996; Stephenson and Kutteh, 2007; The Practice Committee of the American Society for Reproductive Medicine, 2012). The ASRM recommends expectant management as the current standard of care for patients with unexplained RPL (The Practice Committee of the American Society for Reproductive Medicine, 2012). Counseling patients with unexplained RPL to pursue expectant management presents several challenges. Patients often feel an urgency to conceive and expectant management can feel like a passive and time-consuming approach to conception. In addition, patients often carry a significant amount of guilt and grief in association with miscarriage. Attempting spontaneous conception can feel emotionally vulnerable; Despite reassurance of good prognosis, patients doubt that a subsequent pregnancy will be successful (Lachmi-Epstein et al., 2012). For all of these reasons, IVF and preimplantation genetic testing (PGT) have been investigated as a treatment strategy in RPL patients with the goals of shortening time to pregnancy, decreasing CM rates and increasing live birth (LB) rates.

DETAILED DESCRIPTION:
The role of aneuploidy in CM is well known, with over 50% of pregnancy losses attributed to fetal chromosomal abnormalities (Viaggi et al., 2013). Furthermore, for patients greater than 35 years of age with RPL, fetal aneuploidy is responsible for up to 80% of first trimester losses (Marquard et al., 2010). Due to the prevalence of aneuploidy in first trimester losses and in the RPL population, PGT has been proposed as a method for reducing miscarriage by selecting only euploid embryos for transfer (Shahine and Lathi, 2014). The ultimate effect of PGT on increasing LB rates in the RPL population and the time interval to conception are areas of investigation. Current studies are largely retrospective in design with several limitations. For example: Inconsistent definitions of CM and RPL are employed. In addition, the treatment group (IVF and PGT) has been compared with a variety of control groups including IVF without PGT, a control infertile population, or to predicted LB and CM rates based on age and clinical history, but has not been compared with expectant management (Shahine and Lathi, 2014). Finally, the majority of studies report clinical outcomes only of patients who reach PGT biopsy and/or embryo transfer, so all possible cycle outcomes are not captured (Hodes-Wertz et al., 2012).

For the absence of well-designed prospective studies with high level of evidence comparing IVF and PGT to the current standard of care, expectant management, have been performed to date for the treatment of RPL patients. The objective of this study is to perform an intent to treat analysis comparing live birth rate of IVF and PGT to expectant management in fertile RPL patients in one year followed- up period.

ELIGIBILITY:
Inclusion Criteria:

* Age of women <45 years
* Two or more clinical miscarriages with identified foetal chromosomal abnormalities, or three consecutive prior pregnancy losses between 6 and 20 weeks gestational age, excluding biochemical pregnancies.

Exclusion Criteria:

* Presence of APLA including anti-cardiolipin antibody, lupus anticoagulant and b-2-glycoprotein
* Diagnosis for hypothyroidism and hyperprolactinemia with uncontrolled serum thyroid-stimulating hormone and prolactin
* Having a anomaly uterine cavity
* Abormal parental karyotypes (translocation carriers and monogenetic defect)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women who have medical indication attending the Assisted Reproduction clinic, Shanghai First Maternity and Infant Hospital for IVF will be recruited for study after explanation and counseling if they fulfill the inclusion criteria and do not have the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
cumulative live birth rate leading to live birth | 12 Months
  the ongoing status had to be achieved within 12 months since patient inclusion
time to live birth (TTLB). | 24 Months
  TTLB was measured as the time from patient inclusion to a live birth.

SECONDARY OUTCOMES:
Euploidy rate of blastocysts | 30 days
  the number of euploid embryos divided by the total number of blastocysts
Miscarriage rate | 3 months
  the number of miscarriages before 22 weeks per pregnancy
Number of oocytes retrieved | 14 days
  oocytes retrieved per patient
Cycle Cancellation rate | 28 days
  number of PGT cycle with no viable embryo to transfer divided by number of PGT cycle initiated
Clinical pregnancy per transfer /per PGTcycle/per attempt for natural conception | 28 days
  presence of intrauterine gestational sac on ultrasound
Implantation rate | 28 days
  number of gestational sacs per embryo transferred
on-going pregnancy per transfer /per PGTcycle/per attempt | 3 months
  viable pregnancy beyond gestation 8 weeks

OTHER OUTCOMES:
adverse events | 2 years
  : multiple pregnancy, ectopic pregnancy, ,pelvic infection, fetal or congenital defects, obstetric complications, birth weight of babies

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Qin Chen, MD, Principal Investigator — Shanghai first maternty and infant hospital
Locations (1):
- Shanghai first Maternity and Infant health hospital, Tong Ji University, Shanghai, China

REFERENCES:
- [Result] Brigham SA, Conlon C, Farquharson RG. A longitudinal study of pregnancy outcome following idiopathic recurrent miscarriage. Hum Reprod. 1999 Nov;14(11):2868-71. doi: 10.1093/humrep/14.11.2868. PMID 10548638
- [Result] Forman EJ, Hong KH, Ferry KM, Tao X, Taylor D, Levy B, Treff NR, Scott RT Jr. In vitro fertilization with single euploid blastocyst transfer: a randomized controlled trial. Fertil Steril. 2013 Jul;100(1):100-7.e1. doi: 10.1016/j.fertnstert.2013.02.056. Epub 2013 Mar 30. PMID 23548942
- [Result] Lachmi-Epstein A, Mazor M, Bashiri A. [Psychological and mental aspects and "tender loving care" among women with recurrent pregnancy losses]. Harefuah. 2012 Nov;151(11):633-7, 654. Hebrew. PMID 23367735
- [Result] Marquard K, Westphal LM, Milki AA, Lathi RB. Etiology of recurrent pregnancy loss in women over the age of 35 years. Fertil Steril. 2010 Sep;94(4):1473-1477. doi: 10.1016/j.fertnstert.2009.06.041. Epub 2009 Jul 30. PMID 19643401
- [Result] Murugappan G, Ohno MS, Lathi RB. Cost-effectiveness analysis of preimplantation genetic screening and in vitro fertilization versus expectant management in patients with unexplained recurrent pregnancy loss. Fertil Steril. 2015 May;103(5):1215-20. doi: 10.1016/j.fertnstert.2015.02.012. Epub 2015 Mar 13. PMID 25772770
- [Result] Perfetto CO, Murugappan G, Lathi RB. Time to next pregnancy in spontaneous pregnancies versus treatment cycles in fertile patients with recurrent pregnancy loss. Fertil Res Pract. 2015 Apr 21;1:5. doi: 10.1186/2054-7099-1-5. eCollection 2015. PMID 28620510
- [Result] Shahine L, Lathi R. Recurrent pregnancy loss: evaluation and treatment. Obstet Gynecol Clin North Am. 2015 Mar;42(1):117-34. doi: 10.1016/j.ogc.2014.10.002. PMID 25681844
- [Result] Stephenson MD. Frequency of factors associated with habitual abortion in 197 couples. Fertil Steril. 1996 Jul;66(1):24-9. PMID 8752606
- [Result] Stirrat GM. Recurrent miscarriage. Lancet 1990;336:673- 675. The PracticeCommittee of the American Society for ReproductiveMedicine. Evaluation and Treatment of Recurrent Pregnancy Loss: A Committee Opinion. Feril Steril 2012;98:1103 - 1111
- [Result] Regan L, Backos M, Rai R. The Royal College of Obstetricians and Gynaecologists. The RCOG Green-Top Guideline No. 17. The Investigation and Treatment of Couples with Recurrent First-trimester and Second-trimester Miscarriage. 2011
- [Result] Viaggi CD, Cavani S, Malacarne M, Floriddia F, Zerega G, Baldo C, Mogni M, Castagnetta M, Piombo G, Coviello DA, Camandona F, Lijoi D, Insegno W, Traversa M, Pierluigi M. First-trimester euploid miscarriages analysed by array-CGH. J Appl Genet. 2013 Aug;54(3):353-9. doi: 10.1007/s13353-013-0157-x. Epub 2013 Jun 19. PMID 23780398